CLINICAL TRIAL: NCT04099173
Title: A Randomized Pilot Study of a Brief Mindfulness-Based Intervention for Suicidal Ideation
Brief Title: A Brief Mindfulness-Based Intervention for Suicidal Ideation
Acronym: MB-SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00108786
Record Dates: First submitted 2019-07-16; First posted 2019-09-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Suicidal Ideation; Psychiatric Disorder; Addiction
Keywords: mindfulness; suicide related behavior; Veterans; Veterans' Affairs; suicidal ideation
MeSH Terms: conditions — Suicidal Ideation; Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Mindfulness Based Intervention (Experimental): Some participants, as a result of random selection, will be asked to participate in four, 45-minute sessions that will occur on four separate days while on the Inpatient Psychiatric Unit (IPU). These four sessions are in addition to the standard IPU treatment and are experimental. These four sessions will include mindfulness meditation practice and education, creating a Crisis Response Plan, and a brief introduction into self-compassion. As stated above, practicing mindfulness means focusing attention on what is occurring in the present moment in a non-judgmental way. The focus may be on what one is seeing or hearing or physical sensations, such as touch, as well as thoughts and emotions. Meditation is just sitting quietly and practicing mindful awareness.
  Interventions: Behavioral: Brief Mindfulness Based Intervention
- Treatment as Usual (No Intervention): Participants will be asked to fill out several short paper and pencil tests to assess your response to the treatment (10 to 15 minutes) pre-intervention and immediately post-intervention while on the Inpatient Psychiatric Unit (IPU), as well as a follow-up phone call or mail one month after discharge from the IPU. All participants will receive the IPU's normal standard of care treatment (for study purposes this called treatment as usual).

INTERVENTIONS:
Behavioral: Brief Mindfulness Based Intervention — This intervention will consist of four, 45 minute individual mindfulness training sessions (one session per day, over a range of 12 subsequent days) provided by a trained mindfulness facilitator.
  Other Names: MB-SI+ TAU
  Arms: Brief Mindfulness Based Intervention

SUMMARY:
The primary aim of this study is to determine whether a Brief Mindfulness-Based Intervention for Suicidal Ideation (MB-SI) is feasible and safe to implement. The secondary aims are short and longer-term reduction in suicidal ideation (SI) and/or suicide-related behaviors (SRBs) as well as improvements in mindfulness and emotional regulation measures compared to Treatment as Usual (TAU).

DETAILED DESCRIPTION:
The study feasibility will be assessed through participant enrollment and retention numbers. The safety be monitored by the study personnel and include reporting any adverse effects. The intervention fidelity will be aided by standardizing the intervention and ensuring study personnel has the appropriate trainings. Participants will completed questionnaires assessing their SI and SRB as well as mindfulness and emotional regulation measures at three time points (preintervention, immediately postintervention, and 1-month postintervention) and their results will be compared between MB-SI and TAU groups. Additionally, the comparisons will also be conducted for the Emergency Department (ED) admissions, Inpatient Psychiatric Unit (IPU) admissions, and psychiatric ED admissions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with suicidal ideation and any active psychiatric or addictive disorder diagnosis.

Exclusion Criteria:

* Diagnosis of psychotic spectrum illness and current psychotic symptoms or significant cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Measure P1: Change in Columbia Suicide Severity Rating Scale among the MB-SI + TAU cohort compared to the TAU only cohort | pre-intervention and one month post-intervention
  Determine if there is a significant difference in the Columbia Suicide Severity Rating Scale, among the MB-SI + TAU cohort compared to the TAU only cohort. The total Columbia Suicide Severity Rating Scale score can range from 0 to 25, with higher values indicating greater intensity. Longitudinal generalized linear mixed models will be used for the primary analyses. We estimate a total of two time points (baseline and one month follow-up) for the primary outcome.

SECONDARY OUTCOMES:
Measure S1: Number or category of patient and intervention characteristics | throughout the study
  Demographic data extraction will include gender, age, race, ethnicity, religious preferences, service branch, service connection, percent of service connection, diagnosis of psychiatric disorders, substance abuse disorder (SUD) diagnosis, medical diagnosis, and medical diagnosis. In addition, the following factors will also be tracked: the group the participant has been placed in, admission date, consent date, the four intervention dates ( if participant is placed in the treatment group), post-intervention date, and one-month post-intervention date.
Measure S2: Change in psychiatric hospitalizations, emergency room visits for psychiatric illness, and emergency room visits | before the Inpatient Psychiatric Unit (IPU) admission, one-month before the IPU admission, and one-month after the discharge from the IPU
  The change in psychiatric hospitalizations, emergency room visits for psychiatric illness, and emergency room visits, as measured by retrospective review of the electronic medical record, among the MB-SI + TAU cohort will be compared to the TAU only cohort.
Measure S3: Change in TMS among the MB-SI + TAU cohort compared to the TAU only cohort | Pre-intervention, immediately post-intervention, and one month post-intervention
  Determine if there is a significant difference in state or trait mindfulness, as measured by the Toronto Mindfulness Scale (TMS), among the MB-SI + TAU cohort compared to the TAU only cohort. The TMS consists of 2 subscales: curiosity and decentering. Altogether, the TMS includes 13 statements rated on a scale from 0 = not at all, to 4 = very much. Higher values represent higher state of mindfulness.
Measure S4: Change in ERQ among the MB-SI + TAU cohort compared to the TAU only cohort | Pre-intervention and immediately post-intervention
  Determine if there is a significant difference in the Emotional Regulation Questionnaire (ERQ), among the MB-SI + TAU cohort compared to the TAU only cohort. ERQ is a 10-likert-type items designed to measure respondents' tendency to regulate emotions in two ways: cognitive reappraisal and expressive suppression. Scoring is kept continuous and each facet's scoring is kept separate. Higher scores indicate greater capacity for emotional regulation.
Measure S5: Change in Five Facet Mindfulness among the MB-SI + TAU cohort compared to the TAU only cohort | Pre-intervention, immediately post-intervention, and one month post-intervention
  Determine if there is a significant difference in Five Facet Mindfulness among the MB-SI + TAU cohort compared to the TAU only cohort. Five Facet Mindfulness is a scale of 15 items, scores can range from 15 - 75, and higher scores indicate a greater capacity for mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: William R Marchand, MD, LFAPA, Principal Investigator — Salt Lake City Veterans' Administration Medical Center
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herrmann TS, Nazarenko E, Marchand W, Day A, Merrill J, Neil M, Thatcher J, Garland E, Bryan C. Randomized Controlled Trial of a Brief Mindfulness-Based Intervention for Suicidal Ideation Among Veterans. Mil Med. 2024 Feb 27;189(3-4):732-741. doi: 10.1093/milmed/usac291. PMID 36208303